CLINICAL TRIAL: NCT02380911
Title: An Educational Intervention to Improve Effectiveness in the Detection, Treatment and Control of Patients With High Cardiovascular Risk in Low-resource Settings in Argentina: Rationale and Study Design of a Cluster Randomized Controlled Trial.
Brief Title: Statins at the Primary Care Level
Acronym: EPRINA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical Effectiveness and Health Policy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 11526941
Record Dates: First submitted 2015-01-26; First posted 2015-03-05 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Dyslipidemia
Keywords: Dyslipidemia; Global cardiovascular risk; Statins; Educational interventions
MeSH Terms: conditions — Dyslipidemias | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive a multifaceted educational intervention targeting physicians and pharmacist assistants to improve detection, treatment and control of hypercholesterolemia among uninsured patients with moderate-high cardiovascular risk in Argentina.
  Interventions: Other: Educational Intervention
- No Intervention Group (No Intervention): This group will continue with the usual care. Irrespective of the assignment of the clinic to the intervention or control group, all physicians from participating PCCs have received previous training on global cardiovascular risk management, given by the Ministry of Health

INTERVENTIONS:
Other: Educational Intervention — Physicians belonging to the PCC randomized to the intervention group receive a 3-component intervention: education workshop, Educational Outreach Visits and a mHealth application uploaded to their smartphones.
  In addition, 2 intervention support tools are used at the intervention clinics:
  1. A web-based platform that is tailored to send SMS messages for lifestyle modification, and prompts and reminders for clinic appointments are used to improve medication adherence for patients.
  2. On-site training to pharmacist assistants at the first EOV is given by physician trainers focused on counseling to improve medication adherence among patients initiating statin therapy and at each patient visit to the clinic to refill drug prescriptions.
  Arms: Intervention Group

SUMMARY:
Hypercholesterolemia, a major cause of disease burden in both the developed and developing world, is estimated to cause 2.6 million deaths annually (4.5% of all deaths) and one third of ischemic heart diseases., and result in 29.7 million DALY lost. In Argentina, the prevalence of hypercholesterolemia increased between 2005 and 2013 from 27.9% to 29.8%, whereas the rate of non-optimal LDL-C, was 28.0%. The rate of high cholesterol awareness was 37.3 % and the proportion of those who are under pharmacological treatment was dismally low: only 11.1%. Furthermore, only one out of four subjects with a self-reported diagnosis of coronary heart disease (CHD) is taking statins. and most individuals with CHD who are on statins have sub-optimal LDL-C levels. Although other antihypertensive, antidiabetic and low-dose aspirin were available free-of-charge at the primary care clinics of the public sector, statins had not been included until recently. As of 2014, statins (simvastatin 20mg) were incorporated into the package of drugs provided free-of-charge for patients with high cholesterol, according to CVD risk stratification. The goal of this study is to test whether a multifaceted educational intervention targeting physicians and pharmacist assistants, improves detection, treatment and control of hypercholesterolemia among uninsured patients with moderate to high cardiovascular risk in Argentina. Specifically, the intervention will test whether a multifaceted educational intervention program lowers LDL-cholesterol levels and CVD risk in moderate to high cardiovascular risk patients, improves physician compliance with clinical practice guidelines, and improves patient care management and adherence to medication. A cost-effectiveness study will be conducted to compare the intervention to the usual standard of care. This randomized cluster trial will enroll 350 patients from 10 public primary care clinics who will be assigned to receive either the intervention or the usual care. This study is timely and will generate urgently needed data on effective and, practical and sustainable intervention programs aimed at the prevention and control of CVD risk that can be directly used in other primary care settings and health care systems in LMICs.

ELIGIBILITY:
Inclusion Criteria:

* Arteriosclerotic cardiovascular disease: defined as acute coronary syndrome; history of myocardial infarction, stable or unstable angina, coronary revascularization, stroke, or transient ischemic attack presumed to be of atherosclerotic origin and revascularization.
* Moderate-High CVD risk according to the WHO charts adapted by the National MoH (estimated 10-year CVD risk ≥ 20%)
* LDL-C level ≥ 190 mg/dL
* Type 2 diabetes in patients between 40 and 75 years of age

Exclusion Criteria:

* Patients that are already receiving statins, pregnant women, bed-bound, and patients who cannot give informed consent.
* End stage chronics kidney disease receiving dialysis ,HIV/AIDS, tuberculosis, alcohol or drugs abuse.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2015-04; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Cholesterol Level | 1 year
  Net change in LDL-C levels from baseline to month 12 between intervention and usual care groups among all study participants.

SECONDARY OUTCOMES:
Global Cardiovascular Risk | 1 year
  Net change in 10-year-CVD Framingham risk score before and after the implementation of the program.
Clinical practice guidelines compliance | 1 year
  Proportion of patients with high CVD risk who are on statins, and are receiving an appropriate dose according to the CPG.
Cholesterol reduction | 1 year
  Proportion of patients with moderate-high CVD risk who have reduced 30% and 50% of their LDL-C, respectively.
Treatment compliance | 1 year
  Level of treatment adherence evaluated through questionnaire.
Costs of the intervention | 1 year
  Cost-effectiveness of the intervention program.

OTHER OUTCOMES:
Cholesterol Level stratified by history of diabetes | 1 year
  Net change in LDL-C levels from baseline to month 12 between intervention and usual care groups stratified by history of diabetes.
Global Cardiovascular Risk stratified by history of diabetes | 1 year
  Net change in 10-year-CVD Framingham risk score before and after the implementation of the program stratified by history of diabetes.
Clinical practice guidelines compliance stratified by history of diabetes | 1 year
Cholesterol reduction stratified by history of diabetes | 1 year
Treatment compliance stratified by history of diabetes | 1 year
Cholesterol level stratified by 10-year-CVD Framingham risk score level. | 1 year
Clinical practice guidelines compliance stratified by 10-year-CVD Framingham risk score level. | 1 year
Cholesterol reduction stratified by 10-year-CVD Framingham risk score level. | 1 year
Treatment compliance stratified by stratified by 10-year-CVD Framingham risk score level. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo Rubinstein, MD, MSc, PhD, Principal Investigator — Institute for Clinical Effectiveness and Health Policy
Locations (10):
- Argentina (10):
  - Centro de Atención Primaria de la Salud "Dr. Favaloro", Puerto Madryn, Chubut Province
  - Centro de Atención Primaria de la Salud "Ruca Calil", Puerto Madryn, Chubut Province
  - Centro de Atención Primaria de la Salud "Malvinas Argentinas", Rawson, Chubut Province
  - Centro de Atención Primaria de la Salud "Etcheparre", Trelew, Chubut Province
  - Hospital San Luis del Palmar, San Luis del Palmar, Corrientes Province
  - Centro de Atención Primaria de la Salud N°11, Corrientes
  - Centro de Atención Primaria de la Salud Dr. Balbastro, Corrientes
  - Centro de Atención Primaria de la Salud N°13, Corrientes
  - Centro de Atención Primaria "Jardín Residencial", La Rioja
  - Centro de Atención Primaria de la Salud "Faldeo del Velazco", La Rioja

REFERENCES:
- [Derived] Gulayin PE, Lozada A, Beratarrechea A, Gutierrez L, Poggio R, Chaparro RM, Santero M, Masson W, Rubinstein A, Irazola V. An Educational Intervention to Improve Statin Use: Cluster RCT at the Primary Care Level in Argentina. Am J Prev Med. 2019 Jul;57(1):95-105. doi: 10.1016/j.amepre.2019.02.018. Epub 2019 May 23. PMID 31128958
- [Derived] Gulayin P, Irazola V, Lozada A, Chaparro M, Santero M, Gutierrez L, Poggio R, Beratarrechea A, Rubinstein A. Educational intervention to improve effectiveness in treatment and control of patients with high cardiovascular risk in low-resource settings in Argentina: study protocol of a cluster randomised controlled trial. BMJ Open. 2017 Jan 31;7(1):e014420. doi: 10.1136/bmjopen-2016-014420. PMID 28143840